CLINICAL TRIAL: NCT00765453
Title: Randomised Controlled Clinical Trial of the Use of Autologous Bone Marrow Derived Progenitor Cells to Salvage Myocardium in Patients With Acute Anterior Myocardial Infarction
Brief Title: Bone Marrow Derived Adult Stem Cells for Acute Anterior Myocardial Infarction
Acronym: REGEN-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College, London (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Anthony Mathur, Professor, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07/Q0603/76; 2007-002-144
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Heart attack; Anterior Myocardial infarction (MI); adult stem cells; bone marrow progenitor cells; bone marrow stem cells; autologous; left ventricular function; intracoronary injection
MeSH Terms: conditions — Myocardial Infarction; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracoronary (Experimental): Patients will be randomised in a 1:1 ratio to receive intracoronary injections of bone marrow derived stem/progenitor cells or placebo infusion through a percutaneous route
  Interventions: Other: Bone marrow derived progenitor cells or placebo infusion
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Other: Placebo infusion

INTERVENTIONS:
Other: Bone marrow derived progenitor cells or placebo infusion — Over-the-wire balloon catheter delivers infusion into coronary vessel using a stop-flow technique
  Arms: Intracoronary
Other: Placebo infusion — Placebo infusion
  Arms: Placebo

SUMMARY:
Study hypothesis :

The purpose of this study is to determine whether Intracoronary infusion of autologous bone marrow derived progenitor cells to patients undergoing primary angioplasty for acute anterior myocardial infarction will lead to an improvement in cardiac function greater than that seen by placebo alone.

Aims

* To demonstrate that it is safe and feasible to deliver autologous bone marrow derived stem cells within hours of the primary angioplasty procedure
* To demonstrate the effects of autologous bone marrow derived stem cells on cardiac function using cardiac MRI (or cardiac CT), echocardiography and left ventriculography.
* To demonstrate the effect of autologous bone marrow derived stem cells in addition to standard care leads to improvement in cardiac function compared to patients saline(placebo) and standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Heart Attack Centre with acute anterior myocardial infarction (ST elevation in at least 2 contiguous anterior leads ≥ 0.2 mV) and treated with acute PCI with stent implantation within 24 hours after symptom onset
* Acute PCI / stent implantation has been successful (residual stenosis visually < 30% and TIMI flow ≥ 2).
* At the time of inclusion patient no longer requires i.v. catecholamines or mechanical hemodynamic support (aortic balloon pump)
* Significant regional wall motion abnormality in LV angiogram at the time of acute PCI in the LAD territory
* Age 18 - 80 Years (primary angioplasty confers an adverse prognosis in those over the age of 80 years)
* Written informed consent in the recruiting centres native language

Exclusion Criteria:

* Regional wall motion abnormality outside the area involved in the index acute myocardial infarction
* Need to revascularise additional vessels, outside the infarct artery as a planned procedure (these vessels can be treated at baseline)
* Arteriovenous malformations or aneurysms
* Active infection, or fever or diarrhoea within last 4 weeks
* Chronic inflammatory disease
* Known HIV infection or active hepatitis
* Neoplastic disease without documented remission within the past 5 years
* Cerebrovascular insult within 3 months
* Impaired renal function (creatinine > 200mmol) at the time of cell therapy
* Significant liver disease (GOT > 2x upper limit) or spontaneous INR > 1,5)
* Anemia (hemoglobin < 8.5 mg/dl)
* Platelet count < 100.000/µl
* Hypersplenism
* Known allergy or intolerance to clopidogrel, heparin or abciximab
* History of bleeding disorder
* Gastrointestinal bleeding within 3 months
* Major surgical procedure or trauma within 2 months
* Uncontrolled hypertension
* Pregnancy
* Mental retardation leading to inability to obtain informed consent
* Previously performed stem / progenitor cell therapy
* Participation in another clinical trial within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2014-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in left ventricular function (ejection fraction) | 1 year

SECONDARY OUTCOMES:
Longitudinal change in left ventricular function (ejection fraction), change in left ventricular end systolic volume, and change in infarct size | 3 months
Longitudinal change in left ventricular function as measured by LV angiography | 6 months
Longitudinal change in left ventricular function assessed by echocardiography. | 6 months
Change in left ventricular end systolic volume and change in infarct size. | 12 months
Longitudinal change in left ventricular function assessed by echocardiography. | 12 months
MACE | 12 months
Change in Quality of life | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, FRCP FESC Ph, Principal Investigator — Barts and the London NHS Trust
Locations (5):
- Rigshopitalet, Unversity of Copenhagen, Copenhagen, Denmark
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (3):
  - London Chest Hospital, Barts and The London NHS Trust, Bethnal Green, London
  - The Heart Hosptial, UCLH Foundation Trust, London
  - The Royal Free Hospital, Royal Free London Foundation Trust, London

REFERENCES:
- [Derived] Choudry F, Hamshere S, Saunders N, Veerapen J, Bavnbek K, Knight C, Pellerin D, Locca D, Westwood M, Rakhit R, Crake T, Kastrup J, Parmar M, Agrawal S, Jones D, Martin J, Mathur A. A randomized double-blind control study of early intra-coronary autologous bone marrow cell infusion in acute myocardial infarction: the REGENERATE-AMI clinical trialdagger. Eur Heart J. 2016 Jan 14;37(3):256-63. doi: 10.1093/eurheartj/ehv493. Epub 2015 Sep 23. PMID 26405233
- [Derived] Hamshere S, Choudhury T, Jones DA, Locca D, Mills P, Rothman M, Knight C, Parmar M, Agrawal S, Martin J, Mathur A. A randomised double-blind control study of early intracoronary autologous bone marrow cell infusion in acute myocardial infarction (REGENERATE-AMI). BMJ Open. 2014 Feb 18;4(2):e004258. doi: 10.1136/bmjopen-2013-004258. PMID 24549163